CLINICAL TRIAL: NCT05951868
Title: An Innovative Continuum of Care to Promote Exclusive Breastfeeding in Pakistan:a Pilot Randomised Control Trial
Brief Title: An Innovative Continuum of Care to Promote Exclusive Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Health Services Academy, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, zahid azam chaudry, Doctor, Health Services Academy, Islamabad, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2226-HSA
Record Dates: First submitted 2023-06-29; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Breastfeeding
Keywords: exclusive breastfeeding; continuum of care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuum of support on breastfeeding (Experimental): Content of counselling intervention will be on ideal breast feeding practices,benefits of breastfeeding, weaning, myths & common problems faced during breastfeeding with their solutions,Latching techniques,feeding positions, ways to express milk & storage techniques. Discussion and Q&A session
  1. Women with her female family member of support invited for antenatal visit will be counselled by a trained doctor on breastfeeding in 2 -sessions between 32 & 40 weeks of gestation.
  2. Readable booklet & whats app videos having same content in local Urdu language will be shared with the women during antenatal visit and at discharge from hospital.
  3. At time of delivery skin to skin contact, early initiation, proper latching ,positioning and reemphasising on exclusive breastfeeding done by a trained nurse.
  4. Follow up by trained community lady health workers to visit mothers home to reinforce learned information and support mothers at 0,1,2 weeks & 1,3,4,6 months
  Interventions: Behavioral: Continuum of support on breastfeeding.
- Control group/Routine care (No Intervention): The control group will receive routine care in terms of routine counselling done on breastfeeding in the hospital & when mothers at home by lady health workers.

INTERVENTIONS:
Behavioral: Continuum of support on breastfeeding. — A continuous support program for women from antenatal period till 6 months after delivery to initiate early breastfeeding, exclusively breastfeeding for 6 month and to continue breastfeeding till 2 years and beyond.
  Arms: Continuum of support on breastfeeding

SUMMARY:
Malnutrition and non optimal breastfeeding is one the the major cause of high infant morbidity and mortality in a developing country like Pakistan. In addition low women literacy rate,socioeconomic factors, cultural limitations,poor excess to information, misconceptions and other factors has led to low breastfeeding rates.

There has also been a shift over time from home based care and delivery to antenatal care from skilled providers and deliveries within health care facilities. Which is an opportunity to strengthen breastfeeding counselling to mothers starting from health facility where mothers come for antenatal visits and by utilising other modes of counselling within the health facility (which have weak or non-existing structured breast feeding program) and when mothers home till 6 months as a continuous support. Women from different backgrounds have opportunity to get excess to complete information on benefits,misconceptions and myths of breastfeeding which is understandable and acceptable by her, to enable her to make an informed decision to initiate early, exclusively breastfeed and to continue breastfeeding till 2 years or beyond.

The intervention group will receive interventions, will include a family member as a support for participant in her breastfeeding, 2 sessions of counselling on breastfeeding during participants antenatal visits,sharing of readable booklet & video messages on Whats App application of cell phones about breastfeeding, hands on training by nurse after delivery, and continuum of support by multiple visits of lady health workers when the mothers home till 6 months. It will also include training of doctor,nurse & lady health workers involved in the intervention.

The content of intervention will contain benefits & ideal breastfeeding practices, latching & feeding positions,expression & storage of breast milk, associated myths & difficulties with solutions in breastfeeding.

The control group participants will receive the routine support on breastfeeding given in hospital and in the community.

Feasibility, acceptability, cost effectiveness, sustainability and effectiveness of the intervention will be assessed.

DETAILED DESCRIPTION:
Feeding of Infant and young child is a fundamental area to enhance child survival and promote its growth and development As per World Health Organisation (WHO) current global health observatory's data on developing country Pakistan, infant mortality of 53 per 1000 live births and under 5 mortality rate of 63 per 1000 live births is significantly due to malnutrition and non-optimal breast feeding practices.

With a shift to 86% women receiving Antenatal care from a skilled provider, 66% deliveries at health facilities, 69% births attended by skilled providers and 81% percent of births to urban mothers in a health facility..

Also keeping in mind literacy rates, socioeconomic factors, cultural limitations, skills of care providers, limited resource settings, local context, knowledge of mothers on breastfeeding and myths related to breastfeeding, it's an opportunity to initiate and strengthen a continuum of support breastfeeding program starting from hospitals (which have weak or non-existing structured breast feeding program) and extending to community when mothers are at home. In continuum of care program with multi component support interventions starting from antenatal period till 6 months postpartum need to be tested for its feasibility, acceptability, cost effectiveness, sustainability and effectiveness to improve exclusive breast feeding and timely weaning and continued breastfeeding until 2 years or beyond.

After recruitment of 50 women coming for their antenatal checkup as per inclusion/exclusion criteria and by informed consent. Demographic data will be collected and they will be randomly allocated into intervention and control groups.

Care providers involved in the intervention will be trained by a training session.

Intervention group Participants will be invited on next antenatal visits in the health facility;

1. Participants will be accompanied by a female family member of her choice considered as her support ( to encourage and assist mother at home on exclusively breast feeding and continuation of breastfeeding )
2. Participants will be counselled in groups of 5 to 7 in 2 sessions for 45- 60 minutes on benefits & ideal breastfeeding practices, latching & feeding positions, associated myths & difficulties in breastfeeding, discussion and question answer session by a trained doctor in presence of a family member
3. To read Booklet will be given to participants and video recordings having same content as counselling session will be sent by Whats App during antenatal visits and at discharge.
4. At the time of delivery nurse will assist in skin to skin contact, early initiation, proper latching train on feeding positions and reemphasise on exclusive breast feeding.

After delivery and discharge of participant mother from hospital;

1. Trained Lady Health workers (LHWs) of the participant's catchment area will visit at 0,1,2 weeks 1,3,4 & 6 months to reemphasise and support on already learned ideal breastfeeding practices.

The control group participants will receive the routine support on breastfeeding given in hospital and in the community.

Primary & Secondary Outcomes will be measured by a semi structured questionnaire on telephonic call to participants

ELIGIBILITY:
Inclusion Criteria:

1. Age >18years
2. Both nulliparous and multiparous
3. Is between 28-32 week gestation
4. Able to understand and communicate in Urdu/Punjabi
5. Plans her delivery at Aziz Bhatti Shaheed Teaching hospital (ABSTH) Gujrat
6. Has excess to smart phone and Whats App mobile application

Exclusion Criteria:

1. Lady Health Worker currently not present in mothers catchment area.
2. Not able to communicate verbally due to any reason.
3. Known medical conditions, congenital malformations or mental illness that may hinder in breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of interventions | At 7th months after delivery
  The feasibility of the intervention will be assessed through a semi-structured questionnaire administered to all participants and care providers after 6 months of delivery. The questionnaire will evaluate the practicality and ease of implementing the intervention.
Acceptability of interventions | At 7th months after delivery
  The acceptability of the intervention will be determined through a semi-structured questionnaire administered to all participants and care providers after 6 months of delivery. The questionnaire will explore the participants' and providers' satisfaction, comfort, and willingness to continue with the intervention.
Extent to which the intervention is implemented as intended | From enrolment to 7 months
  From enrolment till the last intervention a Performa of every activity ; showing number of participants, day, time, duration, checklist of all the components of intervention delivered and signed by intervention provider on the day of activity with a pictorial evidence sent via Whats App to central record. Feedback from participants on the same checklists of all the components of intervention delivered will also be taken at end of the intervention by an independent researcher.

SECONDARY OUTCOMES:
Infant feeding status | At 2 weeks,1,3 & 6 months after delivery
  Telephonic follow up by research assistant of both intervention and control group mothers with a standard questionnaire using WHO indicators for assessing breastfeeding practices & Survey form of feeding practices at 2 weeks, 1, 3, and 6 months and intentions beyond 6 months
Iowa Infant Feeding Attitude Scale (IIFAS) | After 1 months of delivery
  Telephonic inquiry from participants via translation of Standard adopted 17 question scale form from both intervention and control group
Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | After 3 months of delivery
  Telephonic inquiry from participants via translation of Standard adopted 14-item scale form both intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Zahid A Chaudry, MSPH, Principal Investigator — Department of Gynaecology and Obstetrics teaching unit, Aziz Bhatti Shaheed Teaching Hospital Gujrat
Locations (1):
- Department of Gynaecology and Obstetrics Teaching Unit, Aziz Bhatti Shaheed Teaching hospital (ABSTH), Dhok Gujra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaudry ZA, Naz T, Arshad I, Zahoor A, Javaid M, Sikander S. Innovative continuum of care to promote exclusive breast feeding in Pakistan: protocol of a pilot randomised controlled trial. BMJ Paediatr Open. 2024 May 20;8(1):e002562. doi: 10.1136/bmjpo-2024-002562. PMID 38769049